CLINICAL TRIAL: NCT03439956
Title: Evaluation of Obstetric Outcomes After Transvaginal Specimen Extraction in Gynecological Laparoscopy
Brief Title: Obstetric Outcomes After Transvaginal Specimen Extraction in Gynecological Laparoscopy
Acronym: OUTSET-1
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Università degli Studi dell'Insubria (Other)
Responsible Party: Principal Investigator, Antonio Simone Laganà, Medical Doctor, Università degli Studi dell'Insubria
Other Study IDs: OUTSET-1
Record Dates: First submitted 2018-02-13; First posted 2018-02-20 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Pregnancy Complications; Delivery;Abnormal;Stillbirth
Keywords: Obstetric outcomes; Transvaginal specimen extraction; Gynecological laparoscopy
MeSH Terms: conditions — Pregnancy Complications

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Transvaginal specimen extraction (cases): Pregnant women that underwent previous laparoscopic myomectomy or ovarian cystectomy with transvaginal specimen extraction.
  Interventions: Procedure: Transvaginal specimen extraction
- Controls: Pregnant women that did not undergo previous laparoscopic myomectomy or ovarian cystectomy with transvaginal specimen extraction.

INTERVENTIONS:
Procedure: Transvaginal specimen extraction — Previous transvaginal specimen extraction through posterior colpotomy.
  Groups: Transvaginal specimen extraction (cases)

SUMMARY:
One of the most important downsides of endoscopic surgery is the need to remove surgical specimens of different sizes through very small incisions. This step should ensure the complete retrieval of the surgical specimen with concomitant preservation of its integrity (if possible) in order to avoid intraabdominal contamination of potentially infected or malignant tissues. Possibilities for specimen extraction during laparoscopy include minilaparotomy, enlargement of an ancillary port, transumbilical extraction, and transvaginal extraction through posterior colpotomy.

Although recent evidence has already suggested that transvaginal extraction through posterior colpotomy is a safe and feasible option, to date there are no published data about obstetric outcomes after this procedure.

For this reason, the current study aims to evaluate obstetric outcomes between women that underwent transvaginal specimen extraction through posterior colpotomy and women who did not.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy

Exclusion Criteria:

* Any pre-existent cause of high risk for adverse obstetric outcomes.

Ages: 18 Years to 35 Years | Sex: Female
Age Groups: Adult
Study Population: Pregnant women that underwent previous laparoscopic myomectomy or ovarian cystectomy with transvaginal specimen extraction (cases) and pregnant women that did not.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2023-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Cesarean sections | During the whole study period (2 years).
  Percentage of cesarean sections

SECONDARY OUTCOMES:
Operative deliveries | During the whole study period (2 years).
  Percentage of operative deliveries
Gestational age at deliveries | During the whole study period (2 years).
  Gestational age at the moment of delivery.
Pregnancy complications | During the whole study period (2 years).
  Percentages of complications occurring during pregnancies.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Simone Laganà, M.D., Principal Investigator — Università degli Studi dell'Insubria

IPD SHARING:
Plan to Share IPD: Undecided